CLINICAL TRIAL: NCT06648434
Title: Phase I Trial of MK2 Inhibitor in Combination With mFOLFIRINOX for Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: MK2 Inhibitor in Combination With mFOLFIRINOX for Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202502144; P50CA272213 (NIH)
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; Cancer of the Pancreas
Keywords: Pancreatic cancer; Zunsemetinib; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation phase (zunsemetinib + mFOLFIRNOX) (Experimental): The dose of zunsemetinib will be determined by the dose level assigned and will be taken by mouth either once or twice daily depending on assigned dose level. mFOLFIRINOX will be 85 mg/m^2 of oxaliplatin intravenous (IV) on day 1 of each cycle, 150 mg/m^2 of irinotecan IV on day 1 of each cycle, 400 mg/m^2 of leucovorin IV on day 1 of each cycle, and 2400 mg/m^2 continuous infusion starting on day 1 of each cycle and continuing for 46 hours. Each cycle is 2 weeks in length.
  Interventions: Drug: Zunsemetinib; Drug: mFOLFIRINOX
- Dose expansion phase (zunsemetinib + mFOLFIRNOX) (Experimental): The dose of zunsemetinib will be determined during the dose escalation phase of the trial. mFOLFIRINOX will be 85 mg/m^2 of oxaliplatin intravenous (IV) on day 1 of each cycle, 150 mg/m^2 of irinotecan IV on day 1 of each cycle, 400 mg/m^2 of leucovorin IV on day 1 of each cycle, and 2400 mg/m^2 continuous infusion starting on day 1 of each cycle and continuing for 46 hours. Each cycle is 2 weeks in length.
  Interventions: Drug: Zunsemetinib; Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Zunsemetinib — Patients should take zunsemetinib approximately 12 hours apart (if twice daily dosing) or 24 hours apart (if once daily dosing) at the same time(s) every day, with 8 oz of water.
  Other Names: ATI-450
Drug: mFOLFIRINOX — Includes oxaliplatin, irinotecan, leucovorin, and 5-FU.

SUMMARY:
The investigators hypothesize that MK2 inhibition may improve efficacy of mFOLFIRINOX chemotherapy for patients with pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic ductal adenocarcinoma with no prior systemic treatment for advanced or metastatic disease. Patients with mixed cytology in their tumors such as adeno-squamous, mixed neuroendocrine-carcinoma are permitted if the portion of adenocarcinoma is predominant. Prior adjuvant/neoadjuvant therapy (including FOLFIRINOX or mFOLFIRINOX regimens) is allowed if progression occurred ≥ 12 months from the last dose of that therapy. A biopsy is not required to confirm advanced or metastatic disease.
* Dose escalation: Diagnosis of advanced inoperable or metastatic disease, where mFOLFIRINOX (or classical FOLFIRINOX) is deemed a suitable option per the treating physician.
* Dose expansion: Diagnosis of metastatic disease, where mFOLFIRINOX (or classical FOLFIRINOX) is deemed a suitable option per the treating physician.
* Measurable disease by RECIST 1.1.
* At least 18 years of age
* ECOG performance status ≤ 1.
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm without transfusion within 2 weeks prior to C1D1
  * Hemoglobin ≥ 9.0 g/dL without transfusion within 2 weeks prior to C1D1
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN, unless there are liver metastases in which case AST and ALT ≤ 5.0 x IULN
  * Creatinine clearance > 50 mL/min by Cockcroft-Gault
* Baseline EKG with QTcF ≤ 460 ms.
* Women of childbearing potential and men who are heterosexually active must agree to use adequate contraception as specified in the protocol. Contraception should continue for 1 month following last dose of zunsemetinib, 6 months following last dose of irinotecan, 9 months following last dose of oxaliplatin, and/or 3 months following last dose of fluorouracil. Should a woman (or the female partner of a male participant) become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy with the exception of 1) malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease; 2) or known indolent malignancies that do not require treatment and will likely not alter the course of treatment of metastatic pancreatic cancer.
* History of allogeneic organ or stem cell transplant.
* Currently receiving any other investigational agents, or receipt of an investigational agent within 2 weeks or 5 half-lives of the agent, whichever is shorter.
* Receipt of strong and moderate CYP3A4 and CYP2C8 inhibitors (including grapefruit), strong and moderate CYP3A and CYP2C8 inducers (see Appendices H and I), and drugs with QT prolonging potential within 5 half-lives of cycle 1 day 1.
* Known brain metastases or CNS involvement, because brain metastases are often associated with poor functional status, shortened life expectancy and risk of toxicity.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to zunsemetinib, or other agents used in the study.
* Clinically significant neuropathy ≥ grade 2.
* Presence of interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
* Gastrointestinal conditions which could prevent absorption of zunsemetinib, in the opinion of the treating physician.
* Inability to swallow pills.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia .
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days of C1D1.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Major surgery within 28 days prior to C1D1. Major surgery refers to any surgical procedure that involves general or regional anesthesia, involves extensive resecting or altering of body parts, carries a higher risk of complications, or requires long recovery times. Central line placement is allowed.
* Use of any live vaccines against infectious diseases (eg, influenza, varicella) within 4 weeks (28 days) of C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of zunsemetinib in combination with mFOLFIRINOX (Dose Escalation Only) | Completion of 2 cycles (each cycle is 2 weeks - estimated to be 4 weeks)
Number of participants with dose-limiting toxicities (DLTs) (Dose Escalation only) | Completion of 2 cycles (each cycle is 2 weeks - estimated to be 4 weeks)

SECONDARY OUTCOMES:
Number of participants with adverse events by types | From start of treatment through 30 days after last zunsemetinib dose (estimated to be 13 months)
  Graded by CTCAE v5.
Progression-free rate (PFR) (only for those treated at RP2D) | At 6 months
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and/or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Disease control rate (DCR) (only for those treated at RP2D) | Through completion of treatment (estimated to be 12 months)
  DCR is defined as the number of participants with complete response, partial response, or stable disease) per RECIST 1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and disappearance of all non-target lesions and normalization of tumor marker level.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Overall response rate (ORR) (only for those treated at RP2D) | Through completion of treatment (estimated to be 12 months)
  ORR = defined as number of participants with complete response or partial response by RECIST 1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and disappearance of all non-target lesions and normalization of tumor marker level.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) (only for those treated at RP2D) | Through completion of follow-up (estimated to be 3 years)
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm and/or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Overall survival (OS) (only for those treated at RP2D) | Through completion of follow-up (estimated to be 3 years)
  OS is defined as the duration of time from start of treatment to time of death from any cause.
CA19-9 response rate (only for those treated at RP2D) | Through completion of treatment (estimated to be 12 months)
Change in plasma concentration of zunsemetinib and its metabolites | Cycle 1 day 1 (each cycle is 2 weeks), cycle 2 day 1 (each cycle is 2 weeks), cycle 3 day 1 (each cycle is 2 weeks), cycle 4 day 1 (each cycle is 2 weeks), and end of treatment (estimated to be 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Moh'd Khushman, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who can provide a methodologically sound proposal may direct the proposal to the Principal Investigator at mkhushman@wustl.edu. To gain access, researchers will need to sign a data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu